CLINICAL TRIAL: NCT02277743
Title: A Phase 3 Confirmatory Study Investigating the Efficacy and Safety of Dupilumab Monotherapy Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of Dupilumab Monotherapy Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Acronym: SOLO 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1334
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Experimental): Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection once weekly (qw) from Week 1 to Week 15.
  Interventions: Drug: Placebo (for Dupilumab)
- Dupilumab 300 mg once weekly (qw) (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg every 2 weeks (q2w) (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a placebo alternating with single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Drug: Placebo (for Dupilumab)

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection alternated among the different quadrants of the abdomen, upper thighs and upper arms
  Other Names: REGN668; SAR231893; DUPIXENT®
  Arms: Dupilumab 300 mg every 2 weeks (q2w); Dupilumab 300 mg once weekly (qw)
Drug: Placebo (for Dupilumab) — Subcutaneous injection alternated among the different quadrants of the abdomen, upper thighs and upper arms
  Arms: Dupilumab 300 mg every 2 weeks (q2w); Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group study to confirm the efficacy and safety of Dupilumab monotherapy in adults with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older
2. Chronic AD (according to American Academy of Dermatology Consensus Criteria Eichenfield 2014) that has been present for at least 3 years before the screening visit;
3. Eczema Area and Severity Index (EASI) Score ≥16 at the screening and baseline visits;
4. Investigator's Global Assessment (IGA) Score ≥3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at the screening and baseline visits;
5. ≥10% body surface area (BSA) of AD involvement at the screening and baseline visits;
6. Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable (e.g, because of important side effects or safety risks).

Exclusion Criteria:

1. Participation in a prior Dupilumab clinical study;
2. Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever was longer, before the baseline visit;
3. Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, was likely to require such treatment(s) during the first 4 weeks of study treatment:

   * Immunosuppressive/ immunomodulating drugs (e.g, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.);
   * Phototherapy for AD
4. Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 1 week before the baseline visit;
5. Treatment with biologics as follows:

   * Any cell-depleting agents including but not limited to rituximab: within 6 months before the baseline visit, or until lymphocyte count returns to normal, whichever was longer
   * Other biologics: within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever was longer
6. Regular use (more than 2 visits per week) of a tanning booth/ parlor within 4 weeks of the screening visit;
7. Planned or anticipated use of any prohibited medications and procedures during study treatment;
8. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit;
9. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit. NOTE: Participants might be rescreened after infection resolves;
10. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g, tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per investigator judgment;
11. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening;
12. Positive with hepatitis B surface antigen (HBsAg) or hepatitis C antibody at the screening visit;
13. Participant was a member of the investigational team or his/her immediate family;
14. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study;
15. Women unwilling to use adequate birth control, if of reproductive potential and sexually active.

Note: The information listed above is not intended to contain all considerations relevant to a participant's potential participation in this clinical trial therefore not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (101):
- United States (45):
  - Birmingham, Alabama
  - Fort Smith, Arkansas
  - Rogers, Arkansas
  - Clovis, California
  - Lomita, California
  - Los Angeles, California
  - Oceanside, California
  - Palmdale, California
  - Rolling Hills Estates, California
  - San Diego, California
  - Santa Monica, California
  - Stockton, California
  - Boca Raton, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Newnan, Georgia
  - Chicago, Illinois
  - Normal, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Troy, Michigan
  - St Louis, Missouri
  - Newington, New Hampshire
  - East Windsor, New Jersey
  - Buffalo, New York
  - Corning, New York
  - New Hyde Park, New York
  - Rochester, New York
  - High Point, North Carolina
  - Bethlehem, Pennsylvania
  - Upland, Pennsylvania
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - San Antonio, Texas
  - Waco, Texas
  - Ogden, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Spokane, Washington
- Bulgaria (3):
  - Dupnitsa
  - Plovdiv
  - Sofia
- Canada (8):
  - Winnepeg, Manitoba
  - Bathurst, New Brunswick
  - Hamilton, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Richmond Hill, Ontario
  - Toronto, Ontario
- Denmark (2):
  - Copenhagen
  - Hellerup
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- Germany (12):
  - Berlin
  - Bielefed
  - Blaubeuren Abbey
  - Erlangen
  - Halle
  - Hamburg
  - Hanover
  - München
  - Münster
  - Osnabrück
  - Schwerin
  - Stuttgart
- Japan (19):
  - Kurume, Fukuoka
  - Fukuyama, Hiroshima
  - Inashiki, Ibaraki
  - Yokohama, Kanagawa
  - Habikino, Osaka
  - Neyagawa, Osaka
  - Sakai, Osaka
  - Takatsuki, Osaka
  - Hamamatsu, Shizuoka
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo
  - Nerima-ku, Tokyo
  - Shinagawa, Tokyo
  - Shinjuku, Tokyo
  - Kofu, Yamanashi
  - Gifu
  - Hiroshima
  - Kyoto
  - Osaka
- Singapore, Singapore
- Spain (6):
  - Alcañiz
  - Alicante
  - Barcelona
  - Madrid
  - Seville
  - Valencia

REFERENCES:
- [Result] Simpson EL, Bieber T, Guttman-Yassky E, Beck LA, Blauvelt A, Cork MJ, Silverberg JI, Deleuran M, Kataoka Y, Lacour JP, Kingo K, Worm M, Poulin Y, Wollenberg A, Soo Y, Graham NM, Pirozzi G, Akinlade B, Staudinger H, Mastey V, Eckert L, Gadkari A, Stahl N, Yancopoulos GD, Ardeleanu M; SOLO 1 and SOLO 2 Investigators. Two Phase 3 Trials of Dupilumab versus Placebo in Atopic Dermatitis. N Engl J Med. 2016 Dec 15;375(24):2335-2348. doi: 10.1056/NEJMoa1610020. Epub 2016 Sep 30. PMID 27690741
- [Derived] Langley RG, Gherardi G, Coleman A, Ardeleanu M, Rodriguez-Marco A, Levy S, Bansal A, Chen Z, Rossi AB, Shumel B, Khokhar FA. The Safety Data of Dupilumab for the Treatment of Moderate-to-Severe Atopic Dermatitis in Infants, Children, Adolescents, and Adults. Am J Clin Dermatol. 2025 Nov;26(6):981-1002. doi: 10.1007/s40257-025-00952-w. Epub 2025 Sep 24. PMID 40993471
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Silverberg JI, Lynde CW, Abuabara K, Patruno C, de Benedetto A, Zhang H, Thomas RB, Bego-Le-Bagousse G, Khokhar FA, Vakil J, Marco AR, Levit NA. Efficacy and Safety of Dupilumab Maintained in Adults >/= 60 Years of Age with Moderate-to-Severe Atopic Dermatitis: Analysis of Pooled Data from Four Randomized Clinical Trials. Am J Clin Dermatol. 2023 May;24(3):469-483. doi: 10.1007/s40257-022-00754-4. Epub 2023 Feb 20. PMID 36808602
- [Derived] Paller AS, Silverberg JI, Cork MJ, Guttman-Yassky E, Lockshin B, Irvine AD, Kim MB, Kabashima K, Chen Z, Lu Y, Bansal A, Rossi AB, Shabbir A. Efficacy and Safety of Dupilumab in Patients With Erythrodermic Atopic Dermatitis: A Post Hoc Analysis of 6 Randomized Clinical Trials. JAMA Dermatol. 2023 Mar 1;159(3):255-266. doi: 10.1001/jamadermatol.2022.6192. PMID 36723913
- [Derived] Silverberg JI, Boguniewicz M, Hanifin J, Papp KA, Zhang H, Rossi AB, Levit NA. Dupilumab Treatment in Adults with Moderate-to-Severe Atopic Dermatitis is Efficacious Regardless of Age of Disease Onset: a Post Hoc Analysis of Two Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2731-2746. doi: 10.1007/s13555-022-00822-x. Epub 2022 Oct 21. PMID 36269503
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Armstrong A, Blauvelt A, Simpson EL, Smith CH, Herranz P, Kataoka Y, Seo SJ, Ferrucci SM, Chao J, Chen Z, Rossi AB, Shumel B, Tomondy P. Continued Treatment with Dupilumab is Associated with Improved Efficacy in Adults with Moderate-to-Severe Atopic Dermatitis Not Achieving Optimal Responses with Short-Term Treatment. Dermatol Ther (Heidelb). 2022 Jan;12(1):195-202. doi: 10.1007/s13555-021-00643-4. Epub 2021 Dec 13. PMID 34897582
- [Derived] Paller AS, Tan JKL, Bagel J, Rossi AB, Shumel B, Zhang H, Abramova A. IGAxBSA composite for assessing disease severity and response in patients with atopic dermatitis. Br J Dermatol. 2022 Mar;186(3):496-507. doi: 10.1111/bjd.20872. Epub 2022 Feb 25. PMID 34726270
- [Derived] Griffiths C, de Bruin-Weller M, Deleuran M, Fargnoli MC, Staumont-Salle D, Hong CH, Sanchez-Carazo J, Foley P, Seo SJ, Msihid J, Chen Z, Cyr SL, Rossi AB. Dupilumab in Adults with Moderate-to-Severe Atopic Dermatitis and Prior Use of Systemic Non-Steroidal Immunosuppressants: Analysis of Four Phase 3 Trials. Dermatol Ther (Heidelb). 2021 Aug;11(4):1357-1372. doi: 10.1007/s13555-021-00558-0. Epub 2021 Jun 18. PMID 34142350
- [Derived] Hamilton JD, Harel S, Swanson BN, Brian W, Chen Z, Rice MS, Amin N, Ardeleanu M, Radin A, Shumel B, Ruddy M, Patel N, Pirozzi G, Mannent L, Graham NMH. Dupilumab suppresses type 2 inflammatory biomarkers across multiple atopic, allergic diseases. Clin Exp Allergy. 2021 Jul;51(7):915-931. doi: 10.1111/cea.13954. Epub 2021 Jun 26. PMID 34037993
- [Derived] Boguniewicz M, Beck LA, Sher L, Guttman-Yassky E, Thaci D, Blauvelt A, Worm M, Corren J, Soong W, Lio P, Rossi AB, Lu Y, Chao J, Eckert L, Gadkari A, Hultsch T, Ruddy M, Mannent LP, Graham NMH, Pirozzi G, Chen Z, Ardeleanu M. Dupilumab Improves Asthma and Sinonasal Outcomes in Adults with Moderate to Severe Atopic Dermatitis. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1212-1223.e6. doi: 10.1016/j.jaip.2020.12.059. Epub 2021 Jan 13. PMID 33453450
- [Derived] Silverberg JI, Simpson EL, Guttman-Yassky E, Cork MJ, de Bruin-Weller M, Yosipovitch G, Eckert L, Chen Z, Ardeleanu M, Shumel B, Hultsch T, Rossi AB, Hamilton JD, Orengo JM, Ruddy M, Graham NMH, Pirozzi G, Gadkari A. Dupilumab Significantly Modulates Pain and Discomfort in Patients With Atopic Dermatitis: A Post Hoc Analysis of 5 Randomized Clinical Trials. Dermatitis. 2021 Oct 1;32(1S):S81-S91. doi: 10.1097/DER.0000000000000698. PMID 33165005
- [Derived] Alexis AF, Rendon M, Silverberg JI, Pariser DM, Lockshin B, Griffiths CE, Weisman J, Wollenberg A, Chen Z, Davis JD, Li M, Eckert L, Gadkari A, Shumel B, Rossi AB, Graham NM, Ardeleanu M. Efficacy of Dupilumab in Different Racial Subgroups of Adults With Moderate-to-Severe Atopic Dermatitis in Three Randomized, Placebo-Controlled Phase 3 Trials. J Drugs Dermatol. 2019 Aug 1;18(8):804-813. PMID 31424712
- [Derived] Wollenberg A, Beck LA, Blauvelt A, Simpson EL, Chen Z, Chen Q, Shumel B, Khokhar FA, Hultsch T, Rizova E, Rossi AB, Graham NMH, Pirozzi G, Lu Y, Ardeleanu M. Laboratory safety of dupilumab in moderate-to-severe atopic dermatitis: results from three phase III trials (LIBERTY AD SOLO 1, LIBERTY AD SOLO 2, LIBERTY AD CHRONOS). Br J Dermatol. 2020 May;182(5):1120-1135. doi: 10.1111/bjd.18434. Epub 2019 Dec 1. PMID 31407311
- [Derived] Eichenfield LF, Bieber T, Beck LA, Simpson EL, Thaci D, de Bruin-Weller M, Deleuran M, Silverberg JI, Ferrandiz C, Folster-Holst R, Chen Z, Graham NMH, Pirozzi G, Akinlade B, Yancopoulos GD, Ardeleanu M. Infections in Dupilumab Clinical Trials in Atopic Dermatitis: A Comprehensive Pooled Analysis. Am J Clin Dermatol. 2019 Jun;20(3):443-456. doi: 10.1007/s40257-019-00445-7. PMID 31066001
- [Derived] Silverberg JI, Simpson EL, Ardeleanu M, Thaci D, Barbarot S, Bagel J, Chen Z, Eckert L, Chao J, Korotzer A, Rizova E, Rossi AB, Lu Y, Graham NMH, Hultsch T, Pirozzi G, Akinlade B. Dupilumab provides important clinical benefits to patients with atopic dermatitis who do not achieve clear or almost clear skin according to the Investigator's Global Assessment: a pooled analysis of data from two phase III trials. Br J Dermatol. 2019 Jul;181(1):80-87. doi: 10.1111/bjd.17791. Epub 2019 Apr 11. PMID 30791102
- [Derived] Simpson EL. Dupilumab Improves General Health-Related Quality-of-Life in Patients with Moderate-to-Severe Atopic Dermatitis: Pooled Results from Two Randomized, Controlled Phase 3 Clinical Trials. Dermatol Ther (Heidelb). 2017 Jun;7(2):243-248. doi: 10.1007/s13555-017-0181-6. Epub 2017 May 13. PMID 28503712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 10 countries between 28 Oct 2014 and 12 Feb 2016. A total of 917 participants were screened in the study.
Pre-assignment Details: Out of 917 participants, 671 were randomized and 669 were treated in the study. Participants were randomized in 1:1:1 ratio to receive Dupilumab 300 mg once weekly (qw), Dupilumab 300 mg every 2 weeks (q2w) or Placebo qw.
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a placebo alternating with single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
- Dupilumab 300 mg qw: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab qw from Week 1 to Week 15.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Started | 224 | 224 | 223
Treated | 223 | 223 | 223
Safety Population | 222 (1 participant received at least 1 injection of Dupilumab 300mg(analyzed in Dupilumab 300 mg q2w arm)) | 229 (6 participants (1 [placebo] + 5 [Dupilumab 300 mg qw arm]) analyzed in Dupilumab 300 mg q2w arm) | 218 (5 participants received fewer injections of Dupilumab 300 mg (analyzed in Dupilumab 300 mg q2w arm))
Completed | 184 | 208 | 197
Not Completed | 40 | 16 | 26
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Adverse Event | 10 | 6 | 6
Not completed — Lack of Efficacy | 11 | 4 | 3
Not completed — Other than specified above | 18 | 5 | 16

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw | Total
Number analyzed (Participants) | 224 | 224 | 223 | 671
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.91) | 39.8 (14.68) | 39.3 (14.39) | 39.5 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 94 | 81 | 281
  Male | 118 | 130 | 142 | 390
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 8 | 25
  Not Hispanic or Latino | 212 | 215 | 212 | 639
  Unknown or Not Reported | 1 | 3 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 56 | 54 | 51 | 161
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 10 | 20 | 46
  White | 146 | 155 | 149 | 450
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 3 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  North and South America | 95 | 95 | 96 | 286
  Asia Pacific | 40 | 42 | 38 | 120
  Eastern Europe | 23 | 22 | 24 | 69
  Western Europe | 66 | 65 | 65 | 196
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on scale
    number analyzed (Participants) | 223 | 224 | 223 | 670
    (all) | 34.5 (14.47) | 33 (13.57) | 33.2 (13.98) | 33.6 (14.00)
Investigator's Global Assessment (IGA) Score [Mean (Standard Deviation); unit: units on a scale] — IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0= clear; 1= almost clear; 2= mild; 3= moderate; 4= severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 223 | 224 | 223 | 670
    (all) | 3.5 (0.5) | 3.5 (0.5) | 3.5 (0.5) | 3.5 (0.5)
Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS scale is an assessment tool that is used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0= no itch; 10= worst itch imaginable]). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 224 | 224 | 221 | 669
    (all) | 7.4 (1.77) | 7.2 (1.89) | 7.2 (2.06) | 7.3 (1.91)
Body Surface Area (BSA) Involvement with AD [Mean (Standard Deviation); unit: percentage of body surface area] — Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. Population: Number of participants analyzed = participants with available data for the baseline parameter.
  percentage of body surface area
    number analyzed (Participants) | 223 | 224 | 223 | 670
    (all) | 57.5 (23.38) | 54.7 (23.19) | 56.1 (22.96) | 56.1 (23.17)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: units on a scale] — SCORAD was a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 223 | 223 | 223 | 669
    (all) | 68.3 (13.96) | 66.9 (13.97) | 67.5 (13.61) | 67.6 (13.84)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score indicative of a poor QOL. Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 223 | 224 | 223 | 670
    (all) | 14.8 (7.23) | 13.9 (7.37) | 14.1 (7.51) | 14.2 (7.37)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: units on a scale] — The POEM was a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 223 | 224 | 223 | 670
    (all) | 20.3 (5.90) | 19.8 (6.37) | 20.4 (6.25) | 20.1 (6.17)
Global Individual Signs Score (GISS) [Mean (Standard Deviation); unit: units on a scale] — Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0= none, 1= mild, 2= moderate and 3= severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease). Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 223 | 224 | 223 | 670
    (all) | 9.0 (1.85) | 8.9 (1.81) | 8.9 (1.74) | 9.0 (1.80)
Total Hospital Anxiety Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale] — The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression. Population: Number of participants analyzed = participants with available data for the baseline parameter.
  units on a scale
    number analyzed (Participants) | 204 | 207 | 204 | 615
    (all) | 12.6 (8.33) | 12.2 (7.26) | 12.6 (7.95) | 12.5 (7.85)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Reduction From Baseline of ≥2 Points at Week 16
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing IGA scores at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 224 | 224 | 223
percentage of participants | 10.3 | 37.9 | 37.2
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.7, 95% CI 2-sided [20.18 to 35.17] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.0, 95% CI 2-sided [19.47 to 34.44] — Dupilumab 300 mg qw vs Placebo

2. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment use were set to missing and participants with missing EASI score at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 224 | 224 | 223
percentage of participants | 14.7 | 51.3 | 52.5
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.025 level. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 36.6, 95% CI 2-sided [28.58 to 44.63] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 37.7, 95% CI 2-sided [29.70 to 45.77] — Dupilumab 300 mg qw vs Placebo

3. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were considered as non-responders.
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) included all randomized participants. Here, number of participants analyzed = participants with baseline peak pruritus NRS ≥4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 212 | 213 | 201
percentage of participants | 12.3 | 40.8 | 40.3
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 28.6, 95% CI 2-sided [20.64 to 36.52] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 28.0, 95% CI 2-sided [19.94 to 36.13] — Dupilumab 300 mg qw vs Placebo

4. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥3 Points) of Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥3 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 16 were considered as non-responders.
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) included all randomized participants. Here, number of participants analyzed = participants with baseline peak pruritus NRS ≥3.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 221 | 220 | 211
percentage of participants | 17.2 | 46.8 | 51.7
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous outcome measure was statistically significant); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 29.6, 95% CI 2-sided [21.36 to 37.88] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 34.5, 95% CI 2-sided [26.08 to 42.84] — Dupilumab 300 mg qw vs Placebo

5. Secondary Outcome: Percent Change From Baseline in Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]).
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) included all randomized participants. Here, number of participants analyzed = participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 96 | 169 | 162
percent change | -26.8 (28.38) | -51.1 (28.81) | -49.0 (33.45)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; Least square (LS) mean difference = -24.9, 95% CI 2-sided [-32.26 to -17.52] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -22.8, 95% CI 2-sided [-30.33 to -15.33] — Dupilumab 300 mg qw vs Placebo

6. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 4
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 4 were reported. Values after first rescue treatment were set to missing and subjects with missing peak NRS at Week 4 were considered as non-responders.
Time Frame: Baseline to Week 4
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 212 | 213 | 201
percentage of participants | 6.1 | 16.0 | 23.4
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 9.8, 95% CI 2-sided [3.95 to 15.71] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 17.3, 95% CI 2-sided [10.57 to 23.93] — Dupilumab 300 mg qw vs Placebo

7. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 2
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 2 were reported. Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 2 were considered as non-responders.
Time Frame: Baseline to Week 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 212 | 213 | 201
percentage of participants | 3.3 | 9.4 | 9.5
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0097, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 6.1, 95% CI 2-sided [1.49 to 10.68] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0094, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 6.2, 95% CI 2-sided [1.45 to 10.86] — Dupilumab 300 mg qw vs Placebo

8. Secondary Outcome: Change From Baseline in Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 16
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 96 | 169 | 162
units on a scale | -2.13 (2.044) | -3.78 (2.325) | -3.72 (2.186)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -1.75, 95% CI 2-sided [-2.236 to -1.260] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -1.69, 95% CI 2-sided [-2.189 to -1.186] — Dupilumab 300 mg qw vs Placebo

9. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score to Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 97 | 173 | 162
percent change | -39.5 (33.66) | -73.9 (26.28) | -73.8 (26.41)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -34.6, 95% CI 2-sided [-42.35 to -26.88] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -34.4, 95% CI 2-sided [-42.17 to -26.56] — Dupilumab 300 mg qw vs Placebo

10. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-50 (EASI-50) (≥50% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50 responders were the participants who achieved ≥50% overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment were set to missing and participants with missing EASI-50 scores at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 224 | 224 | 223
percentage of participants | 24.6 | 68.8 | 61.0
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 44.2, 95% CI 2-sided [35.91 to 52.48] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 36.4, 95% CI 2-sided [27.90 to 44.96] — Dupilumab 300 mg qw vs Placebo

11. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-90 (EASI-90) (≥90% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-90 responders were the participants who achieved ≥90% overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment were set to missing and participants with missing EASI-90 scores at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 224 | 224 | 223
percentage of participants | 7.6 | 35.7 | 33.2
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 28.1, 95% CI 2-sided [20.96 to 35.29] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 25.6, 95% CI 2-sided [18.51 to 32.68] — Dupilumab 300 mg qw vs Placebo

12. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) to Week 16
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 97 | 173 | 162
percentage of body surface area | -17.2 (17.381) | -33.72 (19.619) | -35.42 (19.926)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -17.92, 95% CI 2-sided [-22.487 to -13.353] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -18.89, 95% CI 2-sided [-23.125 to -14.650] — Dupilumab 300 mg qw vs Placebo

13. Secondary Outcome: Percent Change From Baseline in the SCORing Atopic Dermatitis (SCORAD) Score to Week 16
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 97 | 172 | 161
percent change | -28.9 (24.25) | -57.2 (24.03) | -56.7 (24.27)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -28.7, 95% CI 2-sided [-35.79 to -21.54] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -28.0, 95% CI 2-sided [-35.09 to -20.87] — Dupilumab 300 mg qw vs Placebo

14. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) to Week 16
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score was indicative of a poor QOL.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 97 | 173 | 162
units on a scale | -5.6 (5.86) | -9.0 (6.61) | -8.8 (6.79)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -4.0, 95% CI 2-sided [-5.16 to -2.80] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -3.7, 95% CI 2-sided [-4.87 to -2.49] — Dupilumab 300 mg qw vs Placebo

15. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) to Week 16
Description: The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 96 | 173 | 162
units on a scale | -5.3 (6.24) | -11.5 (7.07) | -11.3 (6.36)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -6.5, 95% CI 2-sided [-8.02 to -5.01] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -5.9, 95% CI 2-sided [-7.44 to -4.32] — Dupilumab 300 mg qw vs Placebo

16. Secondary Outcome: Change From Baseline in Hospital Anxiety Depression Scale (HADS) to Week 16
Description: HADS is a fourteen item scale. Seven of the items relate to anxiety and seven items relate to depression. Each item on the questionnaire is scored from 0 (minimum score) - 3 (maximum score) and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 82 | 159 | 146
units on a scale | -2.7 (4.40) | -4.8 (5.50) | -4.9 (5.36)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0006, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -2.2, 95% CI 2-sided [-3.44 to -0.95] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -2.2, 95% CI 2-sided [-3.46 to -1.03] — Dupilumab 300 mg qw vs Placebo

17. Secondary Outcome: Percent Change From Baseline in Global Individual Signs Score (GISS) to Week 16
Description: Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0= none, 1= mild, 2= moderate and 3= severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 97 | 173 | 162
percent change | -26.2 (25.70) | -52.5 (27.33) | -51.1 (26.58)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -27.0, 95% CI 2-sided [-35.04 to -18.91] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -25.6, 95% CI 2-sided [-33.06 to -18.12] — Dupilumab 300 mg qw vs Placebo

18. Secondary Outcome: Percent Change From Baseline in Peak Daily Pruritus NRS Score to Week 2
Description: as for outcome 5
Time Frame: Baseline to Week 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 194 | 214 | 212
percent change | -4.2 (22.77) | -20.4 (21.40) | -18.9 (28.40)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg q2w; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -16.5, 95% CI 2-sided [-21.08 to -11.90] — Dupilumab 300 mg q2w vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Dupilumab 300 mg qw; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -15.1, 95% CI 2-sided [-19.62 to -10.50] — Dupilumab 300 mg qw vs Placebo

19. Secondary Outcome: Percentage of Participants With Skin Infection Treatment Emergent Adverse Events (TEAEs) Requiring Systemic Treatment
Description: Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study [Week 28]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. Statistical significance in the hierarchical testing of secondary hypotheses was broken at this endpoint. Therefore, subsequent secondary efficacy endpoints were not tested for statistical significance.
Time Frame: Baseline up to Week 16
Population: Safety analysis set (SAF) which included all randomized participants who received any study drug, and was analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 222 | 229 | 218
percentage of participants | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants With Treatment Emergent Serious Adverse Events (TESAEs) From Baseline Through Week 16
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study [Week 28]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline up to Week 16
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 222 | 229 | 218
percentage of participants | 5.0 | 3.1 | 0.9

21. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Treatment Discontinuation From Baseline Through Week 16
Description: as for outcome 20
Time Frame: Baseline up to Week 16
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 222 | 229 | 218
percentage of participants | 0.9 | 1.7 | 1.8

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 28) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that developed/worsened during the 'on-treatment period' (time form the first dose of study drug up to the end of study [Week 28]). Analysis was performed on safety population.
Groups:
- Placebo: Participants exposed to Placebo (for Dupilumab) for 16 weeks (mean exposure of 14 weeks)
- Dupilumab 300 mg q2w: Participants exposed to Dupilumab 300 mg alternating with placebo qw for 16 weeks (mean exposure of 15 weeks).
- Dupilumab 300 mg qw: Participants exposed to Dupilumab 300 mg qw for 16 weeks (mean exposure of 15 weeks).
Arm/Group | Placebo | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/229 | 0/218
Serious Adverse Events (participants affected / at risk) | 12/222 | 7/229 | 2/218
Other Adverse Events (participants affected / at risk) | 97/222 | 92/229 | 90/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=222) | Dupilumab 300 mg q2w (N=229) | Dupilumab 300 mg qw (N=218)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess sweat gland (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=222) | Dupilumab 300 mg q2w (N=229) | Dupilumab 300 mg qw (N=218)
Conjunctivitis allergic (Eye disorders) | 3 (3) | 12 (13) | 8 (11)
Injection site reaction (General disorders) | 13 (18) | 19 (63) | 41 (111)
Nasopharyngitis (Infections and infestations) | 22 (30) | 27 (32) | 26 (34)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 7 (7) | 12 (14)
Headache (Nervous system disorders) | 13 (16) | 21 (33) | 11 (15)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 66 (77) | 35 (44) | 21 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.